CLINICAL TRIAL: NCT04313478
Title: The Relationship Between Segmental Trunk Control and Gross Motor Performance in Low Birth Weight Born Infant
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 28.03.2014-9
Record Dates: First submitted 2020-03-13; First posted 2020-03-18 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2020-03

CONDITIONS: Early Intervention; Low Birth Weight Infants; Term Infants
Keywords: Early intervention, trunk control, low birth weight, term

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Birth Weight Infants: They were as follows: being at 3 to 9 months' corrected age, gestational age of less than 36 weeks + 6 days, birth weight of 2000 g or less. Infants with any genetic, metabolic, orthopedic congenital abnormalities or chronic diseases and parents' rejection to participate in the study were excluded.
  Interventions: Behavioral: Low Birth Weight and Normal Weight infants
- Normal Weight Infants: They were as follows: being between 3 and 9 months of age, being full-term, had no complications during delivery. Infants that presented any type of sensory or motor disorder were excluded.
  Interventions: Behavioral: Low Birth Weight and Normal Weight infants

INTERVENTIONS:
Behavioral: Low Birth Weight and Normal Weight infants — This cross-sectional study included LBW and NW infants at between 3 and 9 months of age. The levels of trunk control were investigated by using the Segmental Assessment Trunk Control (SATCo). The Alberta Infant Motor Scale (AIMS) were used for assessment of gross motor performance and identify typical and atypical motor development of infants.

SUMMARY:
This study aimed to examine the relation between trunk control and gross motor performance in LBW and NBW infants.

DETAILED DESCRIPTION:
Preterm infants are observed to have reduced trunk extension in the prone position, rigid postural patterns while reaching a toy, fewer movement reactions, trunk rotation, head control, and muscle tone than term infants. To distinguish between the infant with typical motor development and the one with atypical / abnormal motor development and to follow up the level of their trunk controls is important to identify of the motor development delay in the early stage of life.

This cross-sectional study included 42 LBW infants and 43 NBW infants at between 3 and 9 months of age. We investigated the association between the gross motor function and the segmental trunk controls of the LBW infants at the 3-9 months of age compared to NBW infants.

ELIGIBILITY:
Inclusion Criteria:

* the written consent given by the parents,
* being at 3 to 9 months' corrected age,
* gestational age of less than 36 weeks + 6 days,
* birth weight of 2000 g or less.

Exclusion Criteria:

* Infants with any genetic, metabolic, orthopedic congenital abnormalities or chronic diseases and parents' rejection to participate in the study
* Term infants that presented any type of sensory or motor disorder were excluded.

Ages: 3 Months to 9 Months | Sex: All
Age Groups: Child
Study Population: Low birth weight and normal weight infants
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2014-07-30 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Alberta Infant Motor Scale (AIMS) | 15 min
  The gross motor performance of infants were preliminarily evaluated with the Alberta Infant Motor Scale (AIMS). The AIMS, an observational assessment scale, assesses the infants between 0 and 18 months and measures gross motor maturation in infants from birth through independent walking. The AIMS has 58 items, which assess three aspects of motor performance--weight-bearing, posture and antigravity movements in the positions of supine, prone, sitting, and standing positions. A typically developing 18-month-old infant can perform all movements and will obtain a total score of 58. Gross motor performance is defined by the AIMS total score, which is expressed in percentiles based on age. AIMS total score categories were determined by using normative percentile ranges. The categories of gross motor performances were defined as follows: 0-10 atypical development, 11-25 suspected performance, 26-75 normal performance, 76-90 very good performance, 91-100 excellent performance.
Segmental Assessment Trunk Control (SATCo) | 20 min
  The infants were evaluated by using the Segmental Assessment Trunk Control (SATCo). SATCo is the only valid instrument that can assess the level of trunk control by segments and assess the ability of the typical or neuromotor deficient infant to maintain or recover a vertical position while sitting. The infant was positioned in a sitting posture on a wooden bench with the pelvis maintained in a neutral position using a belt system in relation to the vertical axis and with the head upright to identify the level of trunk control. 0 and 1 scores were given according to maintenance of upright posture and the total score was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Seval Kutlutürk, Principal Investigator — Istanbul Medipol University Hospital

IPD SHARING:
Plan to Share IPD: No